CLINICAL TRIAL: NCT01632852
Title: A Phase 1 Study of CSL362 (Anti-IL3Rα / Anti-CD123 Monoclonal Antibody) in Patients With CD123+ Acute Myeloid Leukemia in Complete Remission or Complete Remission With Incomplete Platelet Recovery at High Risk for Early Relapse
Brief Title: A Study of CSL362 in Patients With CD123+ Acute Myeloid Leukemia Currently in Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Limited (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-AML-11-73
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CSL362 (Experimental): See Intervention Description
  Interventions: Biological: CSL362

INTERVENTIONS:
Biological: CSL362 — CSL362 is humanized monoclonal antibody that targets the alpha chain of the interleukin 3 receptor (IL3Rα; also known as CD123) and is optimised for enhanced activation of antibody-dependent cell-mediated cytotoxicity (ADCC) via natural killer cells.
  CSL362 is a sterile solution for injection and will be administered by intravenous infusion to subjects in sequential, escalating dose level cohorts, at doses up to 12.0 mg/kg. CSL362 will be administered every 14 days for a total of 6 infusions per subject. The 6 infusions for each individual subject will contain the same dose of CSL362.

SUMMARY:
This is a first in human, prospective, multicenter, nonrandomized, open-label, dose-escalation study to investigate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of repeat doses of CSL362.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older.
* Previous diagnosis of CD123+ acute myeloid leukemia (AML), de novo or secondary.
* Completed and recovered from all planned induction and consolidation therapy according to the institution's standard of care, and achieved a complete remission (CR)/CR with incomplete platelet recovery (CRp); either first or second CR.
* Has factors conferring high risk of relapse.
* No plans for additional post-remission chemotherapy.
* Not currently a candidate for allogeneic hematopoietic stem cell transplant (HSCT).

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL).
* Known leukemic involvement of the central nervous system.
* Life expectancy 4 months or less as estimated by the investigator.
* Concurrent treatment or planned treatment with other anticancer therapy (chemotherapy, immunotherapy, radiotherapy, targeted therapy, gene therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events (AEs) | From the first treatment (Day 1) up to approximately Day 106
  Number of subjects reporting any AEs and the severity of those AEs.
Dose-limiting toxicity (DLT) evaluation | From the first treatment (Day 1) up to approximately Day 106
  Number of participants with DLT.
  Dose-limiting toxicity (DLT) is defined as:
  * A non-hematological toxicity grade 3 or worse.
  * A hematological toxicity grade 3 that does not recover to baseline within 14 days.
  * A hematological toxicity grade 4 or worse according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.0.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameters | Before each infusion and: at 6 time points within a week after infusion 1, at 1 time point within a week after infusions 2 to 5, at 5 time points within a week after infusion 6, and once at the final visit, approximately 5 weeks after infusion 6
  PK Parameters comprise:
  * Area under the serum concentration time curve (AUC) from time point zero (before dosing):
    * to the time point at which the analyte first returns to baseline (AUC0-last)
    * to a meaningful time after infusion (AUC0-y)
    * extrapolated to infinity (AUC0-∞).
  * The maximum observed serum concentration (Cmax).
  * First time to reach maximum concentration in serum (Tmax).
  * Terminal serum half-life (t 1/2)
Number of subjects developing antibodies against CSL362 | From the first treatment (Day 1) up to approximately Day 106

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mark DeWitte, Study Director — CSL Limited
Locations (5):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University Medical School, Chicago, Illinois
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Weill Cornell Medical College, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Royal Melbourne Hospital, Parkville, Victoria, Australia